CLINICAL TRIAL: NCT03568344
Title: Community Access to Rectal Artesunate for Malaria (CARAMAL): Observational Research in Nigeria, Uganda and DR Congo
Brief Title: Community Access to Rectal Artesunate for Malaria
Acronym: CARAMAL
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: UNITAID (Other); UNICEF (Other); Kinshasa School of Public Health (Other); Akena Associates Ltd. (Unknown); Clinton Health Access Initiative Inc. (Other); Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: P 001-17-1.2
Record Dates: First submitted 2018-05-16; First posted 2018-06-26 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2021-01

CONDITIONS: Malaria
Keywords: Severe malaria; Mortality; Referral; Rectal artesunate; iCCM; Community based treatment
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Community based tx seeking: baseline: Children <5 years of age seeking care for a current/recent febrile illness episode at the level of community based care providers in the study areas, including CHWs and primary health facilities during baseline period (no QA RAS administration).
- tx seeking @ referral facility: baseline: Children <5 years of age seeking care for a severe febrile illness episode directly at the referral facility during baseline period (no QA RAS administration).
- Community based tx seeking: Post RAS: Children <5 years of age seeking care for a current/recent febrile illness episode at the level of community based care providers in the study areas, including CHWs and primary health facilities after QA RAS roll-out (after pre-referral QA RAS administration).
- tx seeking @ referral facility: Post RAS: Children <5 years of age seeking care for a severe febrile illness episode directly at the referral facility after QA RAS roll-out ( no QA RAS administration).

SUMMARY:
Many malaria deaths occur in places where people have poor access to preventive and curative health services. Prompt access to quality health services is critical in the case of severe childhood diseases, among which severe malaria is particularly frequent in endemic areas. In communities where parenteral treatment of severe malaria is not available, the World Health Organization (WHO) recommends administration of a single rectal dose of artesunate (RAS) to children less than 6 years, followed by immediate referral to an appropriate facility where the full package of care for severe malaria can be provided.

Many African countries have already endorsed the use of pre-referral RAS. But treatment guidelines vary widely across these countries and often do not align with the WHO recommendation. With the impending availability of quality-assured rectal artesunate (QA RAS) and countries poised to scale-up this intervention, it is critical to investigate the safe and effective implementation of RAS as part of a continuum of care for severe malaria patients. To ensure that RAS is well targeted, it is equally urgent to learn more about frequency, treatment seeking and risk factors for severe malaria at community level. The CARAMAL project has two major components: the pilot implementation of QA RAS in selected areas of the Democratic Republic of the Congo (DRC), Nigeria and Uganda, and operational research on the introduction of QA RAS into established integrated community case management (iCCM) platforms. The CARAMAL project is funded by Unitaid and coordinated by the Clinton Health Access Initiative, Inc. (CHAI). UNICEF is responsible for QA RAS implementation. Swiss TPH in partnership with the local research organizations Akena Associates Ltd. in Nigeria, Kinshasa School of Public Health in DRC and Makerere University School of Public Health in Uganda carries out the operational research component to generate evidence for the responsible implementation of RAS. Finally, the CARAMAL project will generate a better understanding of severe febrile illness, its management at all levels and key determinants of health outcomes.

DETAILED DESCRIPTION:
Objective(s):

The overall goal of the CARAMAL project is to contribute to reducing malaria mortality in children globally by improving the community management of suspected severe malaria cases. The project will contribute to this goal by advancing the development of operational guidance to catalyse effective and appropriate scale-up of QA RAS as pre-referral treatment of severe malaria.

Accompanying the pilot roll-out of QA RAS by UNICEF, the CARAMAL project will test whether it is feasible to introduce QA RAS into established integrated community case management (iCCM) platforms with only minimal additional supportive interventions and with minimal unintended consequences such as inappropriate use as artemisinin monotherapy.

Through the research activities described in detail below, the CARAMAL project aims to answer the following research questions:

I. What are the minimal requirements of a community case management system to ensure that RAS is an effective part of the continuum of care from the community to a referral facility (defined as a health care facility equipped for inpatient care of severe malaria)?

II. What are the unintended consequences of scaled implementation, such as adverse drug reactions, unforeseen costs [5], or unforeseen issues in treatment of malaria at all levels of care, and how can they be addressed?

III. Is there any use of RAS beyond the recommended guidelines, including full treatment of severe cases with RAS at community level, and the treatment of uncomplicated malaria with RAS?

IV. Can the introduction of pre-referral QA RAS reduce severe malaria case fatality ratio over time under real-world operational circumstances in three distinct settings?

What are the costs and cost-effectiveness of community and peripheral health facility based RAS?

Study Design:

The CARAMAL project has been designed as a multi-country operational research study implemented in three highly malaria-endemic countries. It will be based on a before-and-after plausibility design aligned with the roll-out of QA RAS through established community-based health care provider systems.

Activity 1: A patient surveillance system (PSS) to assess severe febrile illness/suspected severe malaria incidence, case fatality rate, and related clinical patterns, diagnoses, treatment and treatment outcomes from first contact to the point of recovery or death (baseline and after RAS roll-out) Activity 2: Health care provider surveys (HCPS) to establish the availability and uptake of QA RAS at all levels, and health providers' knowledge, attitudes and practices towards RAS (baseline and after RAS roll-out) Activity 3: Household surveys (HHS) to assess treatment seeking, caretakers' knowledge and attitudes towards RAS, and malaria intervention coverage at community level (baseline and after RAS roll-out) Activity 4: An economic evaluation to assess the costs and incremental cost-effectiveness of implementing RAS at community level compared to the current standard of care Activity 5: Routine monitoring of process indicators along the entire case management chain to continuously assess implementation progress of RAS as contextual information for other outcome indicators

Study Population:

Activity 1, Patient surveillance system:

The PSS will include all children <5 years of age seeking care for a current/recent febrile illness episode at the level of community based care providers in the study areas, including Community Health Workers (CHWs) and primary health facilities (HF). All children diagnosed at that level with severe febrile illness / suspected severe malaria will then be enrolled in the PSS and tracked at the referral health facility and at the child's home 28 days after initial diagnosis. In addition, all children <5 years of age seeking care for a severe febrile illness episode directly at the referral facility will be enrolled to evaluate treatment seeking, diagnosis, treatment and disease outcome. These children will be excluded from the case fatality ratio analysis.

Activity 2, Health care provider surveys:

The sampling frame will include all registered providers at all levels operating in the study areas, including public and private providers. A simple random sampling approach stratified by provider level (CHW, primary health facility, etc.) will be used to select providers for the survey.

Activity 3, Household surveys:

Household surveys will include randomly sampled households in the study areas. Households will be selected using a two-stage random sampling approach (village-household) whereas the sampling frames will consist of all villages in the study area and all households in the village, respectively.

In each household, the household heads and parents/caretakers of children < 5 years of age will be eligible to participate.

Measurements and Procedures:

Activity 1, patient surveillance system:

1. CHW / primary health facility (first contact) According to established routine practice, the following procedures are performed: children attending a CHW or primary health facility undergo examination, treatment and referral procedures as per local guidelines. A rapid malaria test (mRDT) is performed on all children with a history of or acute fever, including children with symptoms of severe febrile illness / children with danger signs. The children are then treated as per the applicable national guidelines. Enrolled children will be assigned a unique study ID.
2. Referral facility Children with severe febrile illness / suspected severe malaria and either referred to or directly reporting to a referral facility in the study area will be registered upon arrival in the facility. The study nurse will monitor the case management of each registered patient and continuously enter study-specific details on diagnosis and treatment provided throughout the patient's admission into an electronic case report form.
3. At home (day 28)

   All children with severe febrile illness / suspected severe malaria and enrolled into the patient surveillance system (PSS) by a CHW / primary health facility or at the referral health facility will be followed up at their home by a member of the research team. The primary purpose of this visit is to establish the health status of the child using a structured questionnaire. It will also include a section on the parent's/caretaker's experience and attitude towards the use of RAS. During the home follow-up a finger-prick blood sample will be collected from all of children for:
   * mRDT
   * Microcuvette sample for measuring haemoglobin (Hb) concentration In case of the death of an enrolled child, the research team will attempt to conduct a verbal autopsy at a later stage.

   Activity 2, Health care provider surveys:
4. Health Care Provider Checklist A structured checklist completed to assess the availability of essential medical supplies (incl. RAS) and equipment, human resource capacity, infrastructure and documentation.
5. Health Care Provider Questionnaire An interviewer administered questionnaire with questions pertaining to the health worker's demographics, education and training, work experience and supervision, type and utility of any work-related training received, knowledge, attitudes and practices relevant to febrile case management (incl. diagnostic algorithm and (RAS) treatment guidelines) and intermittent preventive treatment in infants and pregnancy (IPTi, IPTp), experiences implementing malaria/febrile case management and prevention guidelines. More in-depth questions will be asked to health care workers administering RAS as well as different cadres of health workers providing post-referral treatment, focusing on aspects relevant to the implementation of pre-referral RAS and post-referral treatment of severe febrile illness.

Activity 3, Household surveys:

Three survey instruments will be completed with participating household heads and/or household members:

1. Household Questionnaire A structured interviewer administered questionnaire to collect information about coverage and uptake of mosquito nets behaviour change campaigns and other malaria control interventions, alongside background demographic information on each household member as well as indicators of the household's socio-economic status.
2. Treatment Seeking Questionnaire A semi-structured interviewer administered questionnaire completed with randomly selected household members who are parents or caretakers of a child <5 years of age. Parents/caretakers of children who reported a febrile illness (irrespective of severity) in the two weeks prior to the survey will be interviewed about that specific illness episode. The form collects information about the signs and symptoms of the illness and subsequent treatment seeking behaviours, including sources of treatment and types (if any) of drugs administered. Parents/caretakers of children who did not experience a recent febrile illness will be asked about hypothetical care seeking behaviour based on specific vignettes (one scenario of mild and one scenario of severe febrile illness). The form furthermore collects information on the knowledge and attitudes of the parents/caretakers towards RAS. The parent/caretaker will be asked about previous experiences with RAS. Parents/caretakers without any previous experience with RAS will be asked about their attitudes based on a vignette.
3. Prevalence Form / blood sample collection A finger prick blood sample will be taken from every household member below 5 years of age to assess changes in malaria prevalence and anaemia over time in the study areas. A short form will accompany each finger-prick blood sample, recording the individuals' demographic details, recent travel history, intake of any medicine, the mRDT and Hb measurement result, and any treatment administered.

Activity 4, Economic evaluation:

Financial and non-financial economic costs will be collected as part of routine project records over the duration of the study. The evaluation will reflect multiple perspectives including individual (i.e. patient), societal, and health systems-level (i.e. government).

Activity 5, Routine monitoring of process indicators:

Programmatic records of the implementation of QA RAS by UNICEF will be continuously assessed, including:

1. RAS needs assessment data and orders
2. Reports from supportive supervision of CHWs
3. CHW monthly reports
4. CHW, health facility registers

Number of Participants:

Activity 1, Patient surveillance system:

The minimum sample size of 6,032 cases of severe malaria in children < 5 years over 24 months

Activity 2: Health care provider surveys:

* All referral health facilities in the project areas
* All non-referral health facilities in the study area (Uganda and DRC), while in Nigeria, a random sample of 40 facilities will be included.
* 40 community health workers (Nigeria and Uganda).

Activity 3: Household surveys 906 household survey responses on treatment-seeking for severe febrile illness will be required per country and individual survey round.

Study Sites:

* Three health zones in DRC (Kenge, Kingandu and Ipamu),
* A subset of local government areas (LGAs) in one state in Nigeria (Adamawa) , and
* Three districts in Uganda (Apac, Kole and Oyam)

ELIGIBILITY:
Inclusion Criteria:

* Patient surveillance system:
* Children < 5 years
* History of fever plus danger signs indicative of severe febrile illness / suspected severe malaria, according to local iCCM guidelines
* Child referred to higher level facility by CHW/primary health facility, or, child directly attending a referral facility.

Signed full consent form from parent / guardian

Health care provider interview:

* CHW or health worker at peripheral health facility enrolled in the iCCM referral system who treats children < 5 years OR
* Health care provider at referral hospitals treating children < 5 years OR
* Any other health care provider in project area treating children < 5 years
* Signed consent form

Household survey:

* Household head and parent / caregiver of children < 5 years
* Signed consent form from parent / guardian

Exclusion Criteria:

* Patient surveillance system:
* Children ≥ 5 years
* Children with no permanent residence in project area

Health care provider interview:

* Health workers not treating children < 5 years
* Health workers outside project area
* Health workers who do not speak any of the local languages
* Health workers employed since < 1 month

Household survey:

* Parents / guardians with no children < 5 years
* Parents / guardians with no permanent residence in project area
* Parents / guardians who do not speak any of the local languages

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The PSS will include all children <5 years of age seeking care for a current/recent febrile illness episode at the level of community based care providers in the study areas, including CHWs and primary health facilities.
  In addition, all children <5 years of age seeking care for a severe febrile illness episode directly at the referral facility will be enrolled to evaluate treatment seeking, diagnosis, treatment and disease outcome. These children will be excluded from the case fatality ratio analysis.
  During baseline, RAS is expected not to be available at community level in the study area, and the PSS will enroll primarily children not treated with pre-referral RAS, whereas after RAS roll-out, RAS is expected to be administered at the level of community based health care providers.
Sampling Method: Non-Probability Sample
Enrollment: 13758 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of children <5 years with severe febrile illness seen by CHW/primary HF that resulted in death within 28 days | From RAS administration up to 28 days
  Patient surveillance system (data collected at referral facility at 28 days visit including verbal autopsy)

SECONDARY OUTCOMES:
Proportion of children <5 years with severe febrile illness without parasites on day 28 | 28 days after RAS administration
  Rapid diagnostic test for malaria
Proportion of children <5 years with a recent history of fever (mild or severe) who attend CHW/primary HF | Through study completion, an average of 2 years
  Data obtained through Household surveys (semi-structured interviewer administered Treatment Seeking Questionnaire)
Proportion of children <5 years with severe febrile illness seen by CHW/primary HF who completed referral | From RAS administration up to 28 days
  Patient surveillance system (track patients from first point of contact at CHW or primary health facility until referral health facility)
Number of children <5 years with severe febrile illness who report directly to referral health facility | Through study completion, an average of 2 years
  Patient surveillance system (patients with severe febrile illness reporting directly to referral health facility)
Proportion of children <5 years with severe febrile illness managed pre-referral according to guidelines | Through study completion, an average of 2 years
  Patient surveillance system (data collected at CHW / primary HF)
Proportion of children <5 years with severe febrile illness managed post-referral according to guidelines | Through study completion, an average of 2 years
  Patient surveillance system (data collected at referral facility)
Frequency of passively reported adverse events after RAS administration | From RAS administration up to 28 days
  Continuous monitoring of patients medical records (referral facility) for adverse events
Frequency of delayed haemolytic anaemia within 28 days after RAS administration | 28 days after RAS administration
  Hemoglobin measurement
Proportion of trained and functional CHW and primary HF who provide QA RAS | Through study completion, an average of 2 years
  Data obtained through routine monitoring of process indicators along the entire case management chain to continuously assess implementation progress of RAS (Programmatic records)
Proportion of CHW/primary HF with RAS in stock | Through study completion, an average of 2 years
  Data obtained through routine monitoring of process indicators (Programmatic records) and Health care provider surveys (structured checklist to assess the availability of essential medical supplies (incl. RAS) and equipment, human resource capacity, infrastructure and documentation)
Proportion of referral health facilities that have the capacity to manage severe malaria in children in line with global guidance | Through study completion, an average of 2 years
  Data obtained through routine monitoring of process indicators (Programmatic records) and Health care provider surveys (structured checklist to assess the availability of essential medical supplies (incl. RAS) and equipment, human resource capacity, infrastructure and documentation and interviewer administered questionnaires to assess the health worker's demographics, education and training, work experience and supervision, type and utility of any work-related training received, knowledge, attitudes and practices relevant to febrile case management (incl. diagnostic algorithm and (RAS) treatment guidelines) and intermittent preventive treatment in infants and pregnancy (IPTi, IPTp), experiences implementing malaria/febrile case management and prevention guidelines)
Proportion of CHW/primary HF that received at least one supervisory visit in the past 3 months | Through study completion, an average of 2 years
  Data obtained through routine monitoring of process indicators (Programmatic records)
Acceptability of pre-referral RAS among health workers | Through study completion, an average of 2 years
  Qualitative data obtained through Health care provider surveys (interviewer administered questionnaires to assess the health worker's demographics, education and training, work experience and supervision, type and utility of any work-related training received, knowledge, attitudes and practices relevant to febrile case management (incl. diagnostic algorithm and (RAS) treatment guidelines) and intermittent preventive treatment in infants and pregnancy (IPTi, IPTp), experiences implementing malaria/febrile case management and prevention guidelines)
Acceptability of pre-referral RAS among caretakers | Through study completion, an average of 2 years
  Qualitative data obtained through Household surveys (semi-structured interviewer administered Treatment Seeking Questionnaire including attitude towards RAS use)
Total financial cost of managing severe case at community level. Marginal financial cost of adding RAS to the management | From RAS administration up to 28 days
  Costs extracted from the routine accounting documents of the iCCM projects in the three countries, Health care providers surveys and costs incurred by caretakers during referral (PSS Day 28 assessment)
Financial cost of RAS interventions per death averted | Through study completion, an average of 2 years
  Incremental cost-effectiveness of QA RAS introduction over current standard of care for management of severe malaria

CONTACTS AND LOCATIONS:
Overall Officials: Christian Burri, Prof, Principal Investigator — Swiss Tropical & Public Health Institute; Christian Lengeler, Prof, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (3):
- Kinshasa School of Public Health, University of Kinshasa, Kinshasa, Democratic Republic of the Congo
- Akena Associates Ltd., Abuja, Nigeria
- Makerere University School of Public Health, Kampala, Uganda

REFERENCES:
- [Background] Gomes MF, Faiz MA, Gyapong JO, Warsame M, Agbenyega T, Babiker A, Baiden F, Yunus EB, Binka F, Clerk C, Folb P, Hassan R, Hossain MA, Kimbute O, Kitua A, Krishna S, Makasi C, Mensah N, Mrango Z, Olliaro P, Peto R, Peto TJ, Rahman MR, Ribeiro I, Samad R, White NJ; Study 13 Research Group. Pre-referral rectal artesunate to prevent death and disability in severe malaria: a placebo-controlled trial. Lancet. 2009 Feb 14;373(9663):557-66. doi: 10.1016/S0140-6736(08)61734-1. Epub 2008 Dec 6. PMID 19059639
- [Derived] Lengeler C, Burri C, Awor P, Athieno P, Kimera J, Tumukunde G, Angiro I, Tshefu A, Okitawutshu J, Kalenga JC, Omoluabi E, Akano B, Ayodeji K, Okon C, Yusuf O, Brunner NC, Delvento G, Lee T, Lambiris M, Visser T, Napier HG, Cohen JM, Buj V, Signorell A, Hetzel MW; CARAMAL Consortium. Community access to rectal artesunate for malaria (CARAMAL): A large-scale observational implementation study in the Democratic Republic of the Congo, Nigeria and Uganda. PLOS Glob Public Health. 2022 Sep 6;2(9):e0000464. doi: 10.1371/journal.pgph.0000464. eCollection 2022. PMID 36962706
- [Derived] Signorell A, Awor P, Okitawutshu J, Tshefu A, Omoluabi E, Hetzel MW, Athieno P, Kimera J, Tumukunde G, Angiro I, Kalenga JC, Akano BK, Ayodeji K, Okon C, Yusuf O, Delvento G, Lee TT, Brunner NC, Lambiris MJ, Okuma J, Cereghetti N, Buj V, Visser T, Napier HG, Lengeler C, Burri C. Health worker compliance with severe malaria treatment guidelines in the context of implementing pre-referral rectal artesunate in the Democratic Republic of the Congo, Nigeria, and Uganda: An operational study. PLoS Med. 2023 Feb 21;20(2):e1004189. doi: 10.1371/journal.pmed.1004189. eCollection 2023 Feb. PMID 36809247
- [Derived] Hetzel MW, Okitawutshu J, Tshefu A, Omoluabi E, Awor P, Signorell A, Brunner NC, Kalenga JC, Akano BK, Ayodeji K, Okon C, Yusuf O, Athieno P, Kimera J, Tumukunde G, Angiro I, Delvento G, Lee TT, Lambiris MJ, Kwiatkowski M, Cereghetti N, Visser T, Napier HG, Cohen JM, Buj V, Burri C, Lengeler C. Effectiveness of rectal artesunate as pre-referral treatment for severe malaria in children under 5 years of age: a multi-country observational study. BMC Med. 2022 Oct 11;20(1):343. doi: 10.1186/s12916-022-02541-8. PMID 36217159
- [Derived] Brunner NC, Omoluabi E, Awor P, Okitawutshu J, Tshefu Kitoto A, Signorell A, Akano B, Ayodeji K, Okon C, Yusuf O, Athieno P, Kimera J, Tumukunde G, Angiro I, Kalenga JC, Delvento G, Lee TT, Lambiris MJ, Ross A, Cereghetti N, Visser T, Napier HG, Buj V, Burri C, Lengeler C, Hetzel MW. Prereferral rectal artesunate and referral completion among children with suspected severe malaria in the Democratic Republic of the Congo, Nigeria and Uganda. BMJ Glob Health. 2022 May;7(5):e008346. doi: 10.1136/bmjgh-2021-008346. PMID 35580913
- See also: New Unitaid grants help protect women and children from malaria — https://unitaid.org/news-blog/new-unitaid-grants-help-protect-women-and-children-from-malaria/